CLINICAL TRIAL: NCT06147778
Title: Performances and Safety of MuCopilot, a Digital Tool for the Unsupervised Objective Assessment of Cystic Fibrosis
Acronym: MuControl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADS-MuControl-2023
Record Dates: First submitted 2023-10-31; First posted 2023-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MuCopilot comparison to clinical standards (Experimental): Performance of digital tests and questionnaire at Day 0, D1, D3, D5, D7, M1, M2, M3-1 and M3, against clinical standards performed at Day 0 and 3 months.
  Interventions: Device: MuCopilot mobile application

INTERVENTIONS:
Device: MuCopilot mobile application — MuCopilot is a software as medical device with three digital tests, to measure patient's with CF, lung function, global exercise capacity and a questionnaire to address CF symptoms and impacts on some aspects of patient's life

SUMMARY:
The study aims to evaluate MuCopilot, a smartphone application to measure objective data on lung function (cough and dyspnea tests), global exercise capacity (walking test) and patient-reported outcomes (PROs) of patients with Cystic Fibrosis (CF). These data are collected during unsupervised digital tests performed in the patient's home environment between consultations.

The primary objective is to demonstrate the correlation of the MuCopilot digital tests at home (D1) with the results of their standard counterparts (D0) carried out in-clinic.

A secondary objective is to determine the accuracy, reliability and reproducibility of tests results, as well as to study the test-retest of the PRO. The study also aims to assess the safety, usability, and satisfaction of the solution.

Exploratory objectives include evaluating the relationship between MuCopilot's scores and other standards such as FVC, FEV1/FVC ratio as well as to explore the correlation with the cough monitoring with patient's perception.

Patients will be able to download MuCopilot app. They will participate in 1 inclusion visit and 7 follow-up visits, scheduled at Day 1, Day 3, Day 5, Day 7, 1 month, 2 months, 3 months - 1 day.

The study will include 70 CF patients and will be conducted in France.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) patients living with Cystic Fibrosis (CF)
* Enrolled in or benefiting of a Social Security program
* Having read the information sheet and signed the informed consent form
* Owning a personal smartphone which Operating System (OS) is equal or above 14 for iOS (iPhone) and 8 for Android, and have access to a good internet connexion
* Able to read language in which the mobile application is available and able to understand pictograms on the application

Exclusion Criteria:

* History of lung transplantation
* Pregnant women and women who are breastfeeding
* Any medical condition that could interfere with the proper conduct and results of the study (investigator's judgement)
* Illiteracy in French
* Inability to use a smartphone or MuCopilot application
* Persons under legal protection (i.e guardianship or curatorship)
* Participation in another clinical interventional study within 30 days prior to selection or current participation in another study that, in the opinion of the investigator, could interfere with the proper conduct and results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
To demonstrate that the results of the MuCopilot digital tests at home (D1) are associated with the results of their standard counterparts (D0) carried out in-clinic. | During the first in-clinic visit : Day 0 and the first at-home assessment : Day 1
  A correlation coefficient will be used to assess the relationship between MuCopilot tests (MSPT) on Day 1 (at home) and the corresponding standard test on Day 0 (in the clinic). The objective will be achieved if the correlation coefficient reaches a minimum of 0.70. A head-to-head comparison will be performed on the following tests:
  MuCopilot "Mobile Sustained Phonation Test" (MSPT) scores (e.g. maximum phonation time calculated during a sustained phonation assessment) and the FEV1 (air volume exhaled during one second) measured by spirometry at the CF centres
To demonstrate that the results of the MuCopilot digital tests at home (D1) are associated with the results of their standard counterparts (D0) carried out in-clinic. | During the first in-clinic visit : Day 0 and the first at-home assessment : Day 1
  A correlation coefficient will be used to assess the relationship between MuCopilot tests (MEWT) on Day 1 (at home) and the corresponding standard test on Day 0 (in the clinic). The objective will be achieved if the correlation coefficient reaches a minimum of 0.70. A head-to-head comparison will be performed on the following tests:
  MuCopilot "Mobile Endurance Walking Test" (MEWT), i.e. the walking distance (in metres) walked over six minutes on a hard, flat surface at home and the walking distance (in metres) measured during the 6 minute walk test (6MWT) in-clinic

SECONDARY OUTCOMES:
To confirm that the results of the MuCopilot digital test at-home (M3-1) are correlated with their standard clinical counterparts performed in-clinic (M3). | During the last in-clinic visit : at Month 3 and the last at-home assessment Month 3 - 1 day
  According to the same validation principle as for the primaries outcomes, a correlation coefficient will be used to assess the relationship between MuCopilot MSPT and MWT tests at M3 - 1 (at-home) versus standard tests at M3 (in clinic):
  * MuCopilot MSPT scores (sustained phonation time) (at-home) versus Spirometry score FEV1 (air volume exhaled during one second) (in-clinic)
  * MuCopilot MEWT (distance in metres) (at-home) scores versus the 6MWT scores (distance in metres) (in-clinic).
To evaluate the correlation between MuCopilot the digital tests performed in-clinic, and the results of their standard counterparts performed in-clinic | During the first in-clinic visit : Day 0 and the last in-clinic visit : Month 3
  A correlation coefficient will be used to assess the individual correlation between the MuCopilot tests and standard tests performed in-clinic:
  At D0:
  * MSPT scores versus FEV1
  * MEWT scores versus 6MWT At M3
  * MSPT scores versus FEV1
  * MEWT scores versus 6MWT.
To assess intra-patient test-retest reliability of the MuCopilot CF-Scan questionnaire | During at-home visits at Day 1 and Day 3
  Intraclass correlation coefficient (ICC) will be used to assess reliability over time between D1 and D3 (on stable patients without signs or symptoms of CF exacerbation).
  Descriptive analysis of at-home MuCopilot CF-Scan questionnaire between D1 and D3 (Bland-Altman, box plots, etc.).
To assess the safety of the mobile application use. | Throughout the study for all visits in-clinic and at-home Day 0, Day 1, Day 3, Day 5, Day 7, Month 1, Month 2, Month 3-1 day, Month 3
  Adverse events (AEs) and serious adverse events (SAE) related to the use of the application.
To assess the satisfaction and user experience with MuCopilot. | Throughout the study, at-home at Day 7, Month 1, Month 3 - 1 day
  Descriptive analysis of the answers collected in the patient's satisfaction and user experience questionnaires related to the use of MuCopilot.
To assess at-home compliance to MuCopilot. | Throughout the study for all visits in-clinic and at-home Day 0, Day 1, Day 3, Day 5, Day 7, Month 1, Month 2, Month 3-1 day, Month 3
  Descriptive analysis of the number of questionnaires completed or tests performed by patients divided by the number of questionnaires or tests expected by the protocol.
To evaluate the metric performance of the "Mobile Sleep Cough Monitoring Test" (MSCMT) at-home in comparison to ground truth results labelized by specialists. The data will be collected by the mobile application. | Throughout the study for all visits at-home Day 1, Day 3, Day 5, Day 7, Month 1, Month 2, Month 3-1 day and all voluntary tests
  Performance metrics will be used to assess the ability of the digital MSCMT (Mobile Sleep Cough Monitoring Test) trained algorithm to register and automatically detect the cough sounds during sleep to derive :
  * the time spent coughing (in second) : Automatic detection and calculation via MSCMT vs. manual detection and calculcation using annotated data from the mobile application audio record
  * the number of cough : Automatic detection and calculation via MSCMT vs. manual detection and calculation using annotated data from the mobile application audio record.
To evaluate the association between the maximum phonation time determined automatically by the MuCopilot MSPT test at-home and the maximum phonation time evaluated by a trained evaluator on the same dataset. | Throughout the study for all visits at-home Day 1, Day 3, Day 5, Day 7, Month 1, Month 2, Month 3-1 day
  A correlation coefficient will be used to assess the association between the maximum phonation time automatically determined by the MuCopilot MSPT test at-home and the maximum phonation time evaluated by a trained evaluator on the same data (at D1, D3, D5, D7, M1, M2, M3-1).
To evaluate the association between the results of the MSPT and MEWT tests scores in-clinic and the results of these same tests determined by the investigator. | During in-clinic visits at Day 0 and 3 months
  A correlation coefficient will be used to assess the association between the results of the MSPT and MEWT tests scores in-clinic, and the results of these same tests measured simultaneously by the investigator with a stopwatch (time) and an odometer (metres) at D0 and M3.
To assess the reproducibility between MuCopilot tests scores obtained in in-clinic and MuCopilot tests scores obtained at-home | During in-clinic visits at Day 0 and Month 3, and during the at-home visits at Day 1 and Month 3-1 day
  The intraclass correlation coefficient (ICC) will be used to assess the reproducibility of MuCopilot tests MSPT and MEWT performed at :
  * D1 (at-home) versus D0 (in-clinic)
  * M3 -1 (at-home) versus M3 (in-clinic) The minimum ICC to reach is 0.8.
To assess the test-retest reliability of MuCopilot tests scores obtained at-home | During at-home visits at Day 1, Day 3, Day 5 and Day 7
  The intraclass correlation coefficient (ICC) will be used to assess the reliability of MuCopilot tests performed at home at D1, D3, D5 and D7, for MSPT and MEWT digital tests.
  The minimum ICC to reach is 0.8.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Marguet, MD, Principal Investigator — CHU Rouen Charles Nicolle
Locations (7):
- France (7):
  - Centre Hospitalier Lyon Sud (Adultes), Lyon
  - APHM - Hôpital Nord de Marseille, Marseille
  - Centre de compétence Maladies pulmonaires rares Hôpital Pasteur CHU de Nice, Nice
  - American Memorial Hospital, Reims
  - Centre de Perharidy, Fondation Idlys, Roscoff
  - CRCM Mixte - Hôpital Charles Nicolle, Rouen
  - Hôpital Larrey, Toulouse